CLINICAL TRIAL: NCT03418714
Title: Effects of Salvinorin A on Brain Function
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00131537; 5R01DA003889-31 (NIH)
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Drug Effect
MeSH Terms: interventions — salvinorin A

STUDY DESIGN:
Masking Description: Participants will not be aware of exact doses salvinorin A (i.e. they will be told they may receive placebo or up to a moderately high dose of of salvinorin A).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Salvinorin A administration (Experimental): All volunteers will be assigned to the salvinorin A administration arm.
  Interventions: Drug: Salvinorin A

INTERVENTIONS:
Drug: Salvinorin A — Salvinorin A, blinded doses
  Other Names: salvia, salvia divinorum

SUMMARY:
This study will investigate the effects of salvinorin A on human brain activity and connectivity using functional magnetic resonance imaging (fMRI) methods. An inhalation route of administration will be used as it is the most common route for contemporary use of Salvia divinorum, a plant containing salvinorin A.

DETAILED DESCRIPTION:
Volunteers will undergo two experimental sessions that include the inhalation of salvinorin A. The first session will be completed in a comfortable space furnished as a living room, and the second session will be conducted within a magnetic resonance imaging (MRI) scanner.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Have a high school level of education
* Have a history of hallucinogen use and experience with an inhaled psychoactive drug.
* Recent experience (within the past year) with an inhaled psychoactive drug.
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the volunteer does not usually consume caffeinated beverages, he or she must agree not to do so on session days
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages and any tobacco product such as cigarettes or any other nicotine product such as e-cigarettes, within 24 hours of each drug administration. Exceptions include daily use of caffeine.
* Be healthy and psychologically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, and routine medical blood and urinalysis laboratory tests
* Agree that for one week before each session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except if approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals
* Agree not to take any Pro-re-nata (PRN) prescription medications on the mornings of the sessions

Exclusion Criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, or Transient Ischemic Attack (TIA) in the past year
* Seizure disorder or epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking psychoactive prescription medication on a regular (e.g., daily) basis
* More than 25% outside the upper or lower range of ideal body weight
* Current or past history of meeting Diagnostic and Statistical Manual (DSM)-V criteria for schizophrenia, psychotic disorder (unless substance-induced or due to a medical condition), dissociative disorder, bipolar I or II disorder, an eating disorder
* Current or past history of substance-induced psychosis.
* Current or past history within the last 2 years of meeting DSM-5 criteria for moderate or severe alcohol or substance use disorder (excluding caffeine)
* Daily or more frequent tobacco or nicotine use
* Current severe obsessive-compulsive disorder, dysthymic disorder, or panic disorder.
* Current, severe, major depression
* Have a first or second degree relative with schizophrenia, psychotic disorder (unless substance induced or due to a medical condition), or bipolar I or II disorder
* Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to salvinorin A
* Head trauma, traumatic brain injury, or concussion with loss of consciousness for >2 minutes
* Claustrophobia incompatible with MRI scanning
* Medical device incompatible with MRI scanning (e.g. cardiac pacemaker, implanted cardiac defibrillator, aneurysm brain clip, inner ear implant)
* Prior history as a metal worker and/or certain metallic objects in the body -- must complete MRI screening form and be approved by MRI technologist before each scan
* Left-handedness (assessed by the Edinburgh Handedness Inventory)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick S Barrett, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Human psychopharmacology and dose-effects of salvinorin A, a kappa opioid agonist hallucinogen present in the plant Salvia divinorum — https://doi.org/10.1016/j.drugalcdep.2010.11.005

RESULTS

PARTICIPANT FLOW:
Groups:
- Salvinorin A Administration: All volunteers will be assigned to the salvinorin A administration arm.
  Salvinorin A: Salvinorin A (15 micrograms/kg, vaporized), blinded doses
Period: Overall Study
Arm/Group | Salvinorin A Administration
Started | 13
Completed | 12 (One participant moved too much during the practice session and was therefore excluded from the scan.)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Salvinorin A Administration
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.46 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13
Lifetime uses of Salvia divinorum [Mean (Standard Deviation); unit: number of times] — Number of times Salvia divinorum (plant containing salvinorin A) had been used prior to participating in the study.
  number of times | 22.08 (48.70)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Brain Activity (fMRI) as Assessed by Variance in BOLD Signal
Description: Changes in brain activity from before to after salvinorin A administration within canonical brain networks [medial frontal (MF), frontoparietal (FP), default mode (DM), subcortical-cerebellum (SubC), somatosensory-motor (SM), medial visual (MedV), occipital pole (OccP), and lateral visual or (LatV)] will be assessed using blood-oxygenation level dependent (BOLD) techniques. Due to salvinorin A's potential confounding influence on blood flow, activity was assessed by looking at the variance in the BOLD signal. Variance in BOLD signal is a dimensionless variable that can vary from 0 to infinity.
Time Frame: Pre salvinorin A administration and 20 minutes post-salvinorin A administration
Measure: Mean (Standard Deviation); unit: variance in BOLD signal
Arm/Group | Salvinorin A Administration
Number analyzed (Participants) | 12
variance in BOLD signal
  MF activity | 15.65 (74.38)
  FP activity | 18.06 (117.54)
  DM activity | 23.39 (229.30)
  SubC activity | 8.93 (40.91)
  SM activity | 13.06 (79.58)
  MedV activity | 26.15 (406.07)
  OccP activity | 16.96 (366.90)
  LatV activity | 9.30 (77.47)
Statistical Analysis 1: Comparison: Salvinorin A Administration; T test on the change in network activity across all networks, from before to after salvinorin A administration; Test type: Superiority; p = .006, t-test, 2 sided

2. Primary Outcome: Changes in Brain Connectivity (fMRI) as Assessed by Pearson's Correlation
Description: Changes in within and between network functional connectivity (FC) from pre to post-salvinorin A (SA) administration in several brain networks [medial frontal (MF), frontoparietal (FP), default mode (DM), subcortical-cerebellum (SubC), somatosensory-motor (SM), medial visual (MedV), occipital pole (OccP), lateral visual or (LatV)] is assessed via analysis of blood-oxygenation level dependent (BOLD) data. FC is the association between the BOLD activity of two regions over time. This is measured with a Pearson's correlation that is made parametric via z-transformation. FC within a network is the average of all possible pairwise combinations of z-transformed correlations within a network. FC between two networks is the average of all possible pairwise combinations of z-transformed correlations between two networks. We looked at the change in FC from pre to post-SA averaged across participants (this also gives a measure of dispersion).
Time Frame: Pre-salvinorin A administration and 20 minutes post-salvinorin A administration
Measure: Mean (Standard Deviation); unit: Z-transformed Pearson's correlation
Arm/Group | Salvinorin A Administration
Number analyzed (Participants) | 12
Z-transformed Pearson's correlation
  MF within-network connectivity | .01 (.10)
  FP within-network connectivity | .05 (.07)
  DM within-network connectivity | .09 (.06)
  SubC within-network connectivity | .01 (.03)
  SM within-network connectivity | .05 (.09)
  MedV within-network connectivity | .06 (.10)
  OccP within-network connectivity | .05 (.09)
  LatV within-network connectivity | .02 (.08)
  MF-FP between-network connectivity | .02 (.08)
  MF-DM between-network connectivity | .02 (.09)
  MF-SubC between-network connectivity | .00 (.03)
  MF-SM between-network connectivity | .01 (.09)
  MF-MedV between-network connectivity | .01 (.08)
  MF-OccP between-network connectivity | .05 (.10)
  MF-LatV between-network connectivity | .01 (.06)
  FP-DM between-network connectivity | .03 (.05)
  FP-SubC between-network connectivity | .01 (.03)
  FP-SM between-network connectivity | .03 (.08)
  FP-MedV between-network connectivity | .01 (.07)
  FP-OccP between-network connectivity | .04 (.06)
  FP-LatV between-network connectivity | .02 (.05)
  DM-SubC between-network connectivity | .01 (.03)
  DM-SM between-network connectivity | .02 (.06)
  DM-MedV between-network connectivity | .02 (.06)
  DM-OccP between-network connectivity | .02 (.09)
  DM-LatV between-network connectivity | .02 (.06)
  SubC-SM between-network connectivity | .00 (.03)
  SubC-MedV between-network connectivity | .02 (.05)
  SubC-OccP between-network connectivity | .01 (.05)
  SubC-LatV between-network connectivity | .01 (.04)
  SM-MedV between-network connectivity | .02 (.12)
  SM-OccP between-network connectivity | .04 (.10)
  SM-LatV between-network connectivity | .01 (.10)
  MedV-OccP between-network connectivity | .02 (.14)
  MedV-LatV between-network connectivity | .06 (.10)
  OccP-LatV between-network connectivity | .03 (.11)
Statistical Analysis 1: Comparison: Salvinorin A Administration; T test on the change in within- and between-network connectivity across all values, from before to after salvinorin A administration; Test type: Superiority; p = .001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Salvinorin A Administration
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT03418714/Prot_SAP_000.pdf